CLINICAL TRIAL: NCT05872932
Title: Outcome of Combined Botulinum Toxin A Injection and Gastric Balloon Implantation in Obesity Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sebahattin Celik MD (Other)
Responsible Party: Sponsor-Investigator, Sebahattin Celik MD, associate professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-15/03/1374
Record Dates: First submitted 2023-02-19; First posted 2023-05-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: obesity, gastric balloon, botulinum toxin A, intervention
MeSH Terms: conditions — Obesity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Only gastric balloon (Experimental): After analgesia endoscopy will be performed. After diagnostic endoscopy if there is no any gastric pathology that would be contraindication for balloon placement a gastric balloon will be placed. For first day standard medication will be provided. Starting from first hour until 1 week, patient nausea -vomiting and retching scores, re-admission to hospital, quality of life scores will be documented. After analgesia endoscopy will be performed. After diagnostic endoscopy if there is not any gastric pathology that would be contraindication for balloon placement a gastric balloon will be placed. For first day standard medication will be provided. Starting from first hour until 1 week, patient nausea -vomiting and retching scores, re-admission to hospital, quality of life scores will be documented.
  Interventions: Procedure: gastric balloon implantation
- sequential botulinum toxin A injection and then gastric balloon (Experimental): After analgesia endoscopy will be performed. After diagnostic endoscopy if there is not any gastric pathology that would be contraindication for Botox injection and balloon placement, 200 U of botulinum toxin A will be injected to the antrum and the fundus. After 24 hour or 1 week the second procedure (placement of gastric balloon) will be performed. And Starting from first hour until 1 week, patient's nausea-vomiting and retching scores, re-admission to hospital, quality of life scores will be documented.
  Interventions: Procedure: gastric balloon implantation; Procedure: botulinum toxin A injection

INTERVENTIONS:
Procedure: gastric balloon implantation — After diagnostic endoscopy if there is no any gastric pathology that would be contraindication for balloon placement a gastric balloon will be placed
Procedure: botulinum toxin A injection — After diagnostic endoscopy if there is no any gastric pathology that would be contraindication Botox injection and balloon placement, 200 U of Botox A will be injected to antrum and fundus. And 1 week later gastric balloon will be implanted
  Other Names: Gastric balloon implantation 1 week after Botox injection
  Arms: sequential botulinum toxin A injection and then gastric balloon

SUMMARY:
Obesity, which is defined as the accumulation of fat in the body to a degree that impairs health, is defined as a serious public health problem and it is estimated that 13% (approximately 650 million) of the entire world population is obese.

There are different methods in the fight against obesity, one of these methods is bariatric interventions. Although bariatric surgery is the most effective of these procedures, the tendency to endoscopic methods is increasing due to the surgical risk. Gastric balloon is the most common endoscopic method. In addition, gastric botox is among the methods used.

Health consequences of endoscopic interventions have been widely investigating and while gastric balloon recommended as safe and effective method, the situation for gastric botox is controversial.

Although it seems as gastric balloon is an office procedure and safely performed, especially the first week is difficult process for patients. It can also end with abdominal pain, nausea, retching, and eventually a process leading to premature removal of the balloon. In Italian study, Genco et al. reported that out of 2515 patients 11 patients (0.44%) balloon removed due to psychological intolerance. While the reported rate of early gastric balloon removal generally ranges from 0.44% to 16%, De Castro ML. et al. reported the early removal rate as 20%. While the complications related to the gastric balloon are as stated, problems such as nausea, vomiting and cramps after the gastric botox procedure are either not reported or not seen at all.

Therefore, we hypothesize that sequential endoscopic procedures (first botox application followed by gastric balloon placement) will reduce these early complications (abdominal pain, nausea, retching) and early removal of the gastric balloon.

The only study we have reached regarding combined therapy was done in Turkey. Kanlıöz M et al. reported that combining botox and balloon was found to be more effective in losing weight, but it was stated that it had more side effects. In this study, we think that the side effects may already be related to the balloon. As James A et al. stated in their experimental work, the effectiveness of botox is time dependent. It has been stated that the efficacy is optimal after 6 hours in injections to the pyloric region.The fact that the balloon was inserted in the same session, without waiting for enough time after the botox procedure to be effective, may have reduced the possible protective effect of the botox.

ELIGIBILITY:
Inclusion Criteria:

1. patients with body mass index over 30
2. patients who have been on a diet and have done sports at least for 6 month and yet could not lose weight.
3. 18-65 years old patients

Exclusion Criteria:

1. patients diagnosed with peptic ulcer
2. untraceable patients after injection of botulinum toxin A
3. patients with no history of bariatric surgery or interventions
4. patients who do not retrieve balloon after 6 month or require repetitive implantations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop intolerance and undergo balloon removal procedure | First 6 months after intragastric balloon placement
  Number of patients who develop intolerance and undergo balloon removal procedure
Quality of life measured using SF-36 questionnaire | The questionnaire will be taken 1 week after the balloon placement
  The acute(1 week) time frame format of Short Form-36 questionnaire will be used to assess health-related quality of life
Nausea-vomiting and retching measured using Rhodes index of nausea-vomiting-retching(RİNVR) | The questionnaire will be taken 6 hours after intragastric balloon placement
Number of analgesics and muscle relaxants needed | First week after intragastric balloon placement
Weight loss | 6 months after intragastric balloon placement

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University Faculty of Medicine, Van, Turkey (Türkiye)